CLINICAL TRIAL: NCT00173862
Title: A Phase II Study of Gemcitabine and Ifosfamide As a Second-Line Systemic Chemotherapy for Cisplatin -Failed Advanced Transitional Cell Carcinoma
Brief Title: Gemcitabine and Ifosfamide As a Second-Line Systemic Chemotherapy for Cisplatin -Failed Advanced TCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 155I1
Record Dates: First submitted 2005-06-30; First posted 2005-09-15 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2005-06

CONDITIONS: Transitional Cell Carcinoma
Keywords: Combination, Chemotherapy,transitional cell carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Gemcitabine; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Gemcitabine, Ifosfamide

INTERVENTIONS:
Drug: Gemcitabine, Ifosfamide

SUMMARY:
The purpose of this study is to evaluate the efficacy of Gemcitabine plus Ifosfamind as second line chemotherapy in advanced transitional cell carcinoma in terms of response rate and overall survival .

DETAILED DESCRIPTION:
Cisplatin-based combination chemotherapy produces a response rate of 40-70% in TCC patients. However, only less than 10% of the patients can achieve long-term remission. Until now, there is no standard chemotherapy for cisplatin-failed TCC patients. Both gemcitabine and ifosfamide have been identified to have response rates of 20% or more in pretreated TCC patients. It is thus reasonable to combine these two active drugs as a second-line treatment for TCC.

Patients enrolled must have a pathologically proven urothelial transitional cell carcinoma (TCC) and must have exposed to one cisplatin-based combination chemotherapy for the advanced disease. GI regimen will be continued until maximal response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed transitional cell carcinoma
* Advanced / metastatic disease failed to prior chemotherapy (diagnostically confirmed disease progression during the treatment of last chemotherapy or within 6 months after the end of last chemotherapy)
* Presence of at least one measurable disease which is defined as lesion that can be measured in at least 1 dimension as ³ 20 mm with conventional technique or ³ 10 mm with spiral CT scan
* Performance status of ECOG 0, 1, 2
* Age 20 years or older
* Life expectancy more than 3 months
* Adequate hematopoietic function as defined below:

  * WBC ³ 3,000/uL
  * Platelets ³ 75,000/Ul
* Adequate organ function as defined below:

  * Total bilirubin £ 1.5 ´ ULN
  * ALT / AST£ 5 ´ ULN
  * Creatinine £ 1.5 mg/dL
* Adequate serum electrolyte concentration:

  * 4 mmol/L<[K+] <5.3 mmol/L
  * 0.74 mmol/L<[Mg2+] <1.03 mmol/
  * 2.02 mmol/L<[Ca2+]<2.60 mmol/L
* Result of ECG assessment: QTC < 460 msec
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Received chemotherapy, radiotherapy, surgery, or other investigational drug within 4weeks prior to entering the study
* Receiving other concurrent palliative chemotherapy, radiotherapy, hormonal therapy, or other investigational drug except non-disease related conditions (e.g. insulin for diabetes) during study period
* Presence of CNS metastasis
* Previous or current malignancy with the exception of curatively treated non- melanoma skin cancer or cervical carcinoma in situ
* Presence of serious concomitant illness which might be aggravated by study medication:

  1. Uncontrolled infection (active serious infections that are not controlled by antibiotics)
  2. Peripheral neuropathy grade 2 or higher (by NCI common toxicity criteria in sensory or motor neuropathy)
  3. Clinically significant arrhythmia (electrocardiogram QTc greater than 500 msec)
  4. Prior myocardial infarction or serious coronary arterial disease within the last 12 months
* Mental status is not fit for clinical trial.
* Women of child-bearing potential (pregnancy or breast feeding)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2000-05; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Response rate | 2000~2006

SECONDARY OUTCOMES:
Overall Survival, Safety | 2000~2006

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hung Hsu, M.D., Ph.D., Principal Investigator — Department of Oncology , National Taiwan University Hospital; Ann-Lii Cheng, M.D., Ph.D., Study Chair — Department of Oncology, National Taiwan University Hospital
Locations (1):
- Department of Oncology , National Taiwan University Hospital, Taipei, Taiwan